CLINICAL TRIAL: NCT06388772
Title: Phase I Clinical Study of Tolerability, Safety and Pharmacokinetics of QHRD106 Injection in Chinese Healthy Subjects With Single Doses
Brief Title: Study to Assess PK, Safety and Tolerability Early in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Changzhou Qianhong Bio-pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HJG-CZQH-QHRD106
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part-A SAD in healthy subjects(Cohort 1-8) (Experimental): A randomized, double-blinded, placebo-controlled, single ascending dose (SAD) study in healthy male and female subjects. Subjects will receive QHRD106 by intramuscular-injection (im).
  Interventions: Drug: QHRD106 Injection
- Part-B Healthy subjects SAD placebo (Experimental): A randomized, double-blinded, placebo-controlled, single ascending dose (SAD) study in healthy male and female subjects. Subjects will receive placebo by intramuscular-injection (im).
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: QHRD106 Injection — 250IU~8400IU,pegylated(PEG)-tissue kallikrein-1
  Other Names: pegylated(PEG)-tissue kallikrein-1
  Arms: Part-A SAD in healthy subjects(Cohort 1-8)
Drug: placebo — placebo
  Arms: Part-B Healthy subjects SAD placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics (PK) of QHRD106 early in Chinese healthy subjects with single doses.

DETAILED DESCRIPTION:
Eight dose groups were initially set up. The experimental groups were increased from low to high dose according to the principle of increasing dose, and Placebo was added as the control group. All the selected subjects in the experimental group were given the drug once.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects, male and female equally;
2. Aged between 18 and 50 at the time of screening (including boundary values); Male weight ≥50.0kg, female weight ≥45.0kg; All subjects had a body mass index (BMI) between 19 and 28kg/m2 (including boundary values);
3. Participate voluntarily and sign informed consent to complete the experiment according to the research protocol.

Exclusion Criteria:

Subjects who meet one of the following conditions will not be enrolled in the trial:

1. a person who is allergic to, or is allergic to, 2 or more drugs or foods, or is known to have a history of allergy to the test preparation and any of its components or related preparations;
2. Patients with a history of clinically serious diseases such as nervous system, blood circulatory system, digestive system, urinary system, respiratory system, immune system, endocrine system, malignant tumor, mental and metabolic abnormalities, or any clinically significant diseases judged by researchers to be in an active period or unstable state;
3. Based on vital signs (including sitting blood pressure, pulse, and body temperature), physical examination, 12-lead electrocardiogram examination, and laboratory examination (including routine blood routine, urine routine, blood biochemistry, and coagulation function), the investigator determined that the abnormality was clinically significant;
4. postural hypotension;
5. α1-antitrypsin deficiency;
6. Patients with difficulty in venous blood collection;
7. People with a history of fainting needles and fainting blood;
8. A history of drug abuse within the last two years (including repeated and heavy use of various narcotic drugs and psychotropic substances for non-medical purposes);
9. Excessive smoking within 3 months before screening (average > 5 cigarettes/day) or unable to stop using any tobacco products during the test period or smokers within 48 hours before screening;
10. Excessive daily consumption of tea, coffee or caffeinated beverages (more than 8 cups per day, 1 cup =250mL) in the 3 months before screening;
11. alcoholics (i.e. men drinking more than 28 standard units per week, women drinking more than 21 standard units per week, 1 standard unit containing 14g of alcohol, such as 360mL beer or 45mL spirits with 40% alcohol or 150mL wine) or regular drinkers (i.e. more than 14 standard units per week) in the six months prior to screening;
12. Positive alcohol breath test (test result greater than 0.0mg/100mL);
13. Hepatitis B surface antigen (HBsAg), hepatitis C virus(HCV) antibody, syphilis antibody and human immunodeficiency virus(HIV) antibody test one or more positive;
14. Positive urine screening for drug abuse (including morphine, methamphetamine, ketamine, dimethylene dexamphetamine, tetrahydrocannabinol, cocaine);
15. Abnormal chest X-ray or CT findings with clinical significance;
16. Abdominal B-ultrasonography (liver, bile, pancreas, spleen and kidney) with abnormal results and clinical significance;
17. Severe acute bacterial, viral or fungal infection within 4 weeks prior to screening;
18. Patients who had used any protease drugs (such as chylase, indinavir sulfate, ritonavir, bortezomib, ixazomib citrate, etc.) within 4 weeks before screening;
19. Use of any prescription or over-the-counter drugs, as well as any functional vitamins or Chinese herbal products within 2 weeks prior to screening;
20. Blood donation or blood loss greater than 400mL within 3 months before screening (except physiological blood loss);
21. Vaccinated within 1 month before screening, or planned to be vaccinated during the study period and within 1 month after the study ends;
22. Those who had undergone surgery within 3 months prior to screening or planned to undergo surgery during the trial;
23. Participants who participated in any drug clinical trial as a subject within 3 months before enrollment;
24. have consumed a special diet (including grapefruit, chocolate, tea, cola, or any food or beverage containing caffeine, alcoholic beverage, or other food or beverage that affects the absorption, distribution, metabolism, or excretion of drugs) in the 48 hours prior to screening;
25. The subjects or their partners do not wish to use one or more non-drug contraceptive methods (such as total abstinence, condoms,contraceptive rings, ligation, etc.) for contraception during the trial period or have pregnancy plans within 3 months after the end of the study; Or screening women with positive pregnancy tests or breastfeeding women;
26. With magnetic resonance examination contraindications: metal implant, claustrophobia, etc.;
27. Other situations in which the investigator considers that participation in the trial may not be appropriate. -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by incidence, severity, and causality of adverse events | Up to 36 days after final dose
  The frequency and number of adverse events, adverse reactions and serious adverse
Plasma measurements of QHRD106 | Up to 36 days after final dose
  The concentration of a single dose was measured at 8 different doses

CONTACTS AND LOCATIONS:
Overall Officials: Juan Li, Doctor, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang L, Sun R, Song H, Chen Z, Hong Y, Yang H, Zhang Y, Wei L, Fei F, Li J. The first-in-human study of QHRD106 functioning as a safe and effective long-acting kallikrein drug potentially aiding ischemic stroke. Expert Opin Investig Drugs. 2024 Dec;33(12):1257-1265. doi: 10.1080/13543784.2024.2430200. Epub 2024 Nov 19. PMID 39545461